CLINICAL TRIAL: NCT01156883
Title: Young Adult Acute Lymphoid Leukemia (ALL): Intensification of Pediatric AIEOP LLA-2000 Treatment
Brief Title: Combination Chemotherapy in Treating Young Adult Patients With Acute Lymphoblastic Leukemia
Acronym: LAL1308
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1308; GIMEMA-LAL1308; EU-21042
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Leukemia
Keywords: B-cell adult acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Ifosfamide; Mercaptopurine; Methotrexate; Methylprednisolone; Prednisone; Thioguanine; Vincristine; Vindesine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Drug: mercaptopurine
Drug: methotrexate
Drug: methylprednisolone
Drug: prednisone
Drug: thioguanine
Drug: vincristine sulfate
Drug: vindesine

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with steroid therapy may kill more cancer cells.

PURPOSE: This clinical trial is studying the side effects of combination chemotherapy in treating young adult patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility of combination chemotherapy in young adult patients with acute lymphoid leukemia.
* To determine the complete response rate at the end of induction therapy in these patients.
* To determine the overall survival of patients treated with these regimens.
* To determine the disease-free survival of patients treated with these regimens.
* To determine the event-free survival of patients treated with these regimens.
* To determine toxicity of these regimens.
* To determine compliance related to dose intensity.

OUTLINE:

* Steroids prephase therapy: All patients receive steroids (i.e., prednisone or methylprednisolone) and methotrexate.
* Induction therapy (induction Ia followed by Ib): Patients receive induction Ia comprising vincristine, daunorubicin hydrochloride, asparaginase, and prednisone. They then receive induction Ib comprising cyclophosphamide, mercaptopurine, and cytarabine. Patients who achieve hematological remission proceed to consolidation therapy.
* Consolidation therapy: Patients receive consolidation therapy according to risk group.

  * Standard-risk patients: Patients receive high-dose methotrexate and mercaptopurine.
  * High-risk patients: Patients receive consolidation therapy in 3 steps.

    * Step 1: Patients receive dexamethasone, vincristine, methotrexate, cytarabine, and asparaginase.
    * Step 2: Patients receive dexamethasone, vindesine, methotrexate, ifosfamide, asparaginase, and daunorubicin hydrochloride.
    * Step 3: Patients receive dexamethasone, cytarabine, and asparaginase. After completion of consolidation therapy, patients proceed to reinduction therapy.
* Reinduction therapy (reinduction IIa followed by IIb): Patients receive reinduction IIa comprising vincristine, doxorubicin hydrochloride, asparaginase, and dexamethasone. Patients then receive reinduction IIb comprising cyclophosphamide, thioguanine, and cytarabine.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoid leukemia, meeting any of the following criteria:

  * Non-mature B-cell disease
  * Non-Philadelphia chromosome positive disease
  * T -cell or B-cell phenotype

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Prior pretreatment with antiblastic chemotherapy allowed

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2010-04; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Treatment feasibility | At 24 months from study entry.
  To determinate if the Risk-adapted, MRD-directed therapy improves the estimation of Overall Survival (OS) at 24 months from study entry.

SECONDARY OUTCOMES:
Disease free survival | At three years from study entry
  Estimation of Disease Free Survival (DFS).
Event free survival | At 3 years from study entry
  Estimation of Event Free Survival (EFS).
Overal survival | At 3 years from study entry
Safety | At 3 years from study entry
  Grade III-IV toxicity events
Compliance | At 3 years from study entry
  Therapy compliance

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foa, MD, Principal Investigator — Universita Degli Studi "La Sapeinza"
Locations (43):
- Italy (43):
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma, (RM)
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - USL 8 - Ospedale S.Donato, Arezzo
  - Dipartimento Area Medica - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - UO Ematologia con trapianto- AOU Policlinico Consorziale di Bari, Bari
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia e Fisiopatologia delle Emostasi - Azienda Ospedaliera - Arcispedale S. Anna, Ferrara
  - Divisione Ematologia 1 - Azienda Ospedaliera Universitaria "San Martino", Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Ospedale Niguarda " Ca Granda", Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - UOSC di Ematologia Oncologica - Istituto Nazionale Tumori "Fondazione Senatore Giovanni Pascale", Napoli
  - zienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Inferiore U.O. Medicina Interna Ematologia ed Oncologia P.O. Umberto I, Nocera Inferiore
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Divisione di Ematologia - Ospedale S. Camillo Divisione di Ematologia - Ospedale S. Camillo, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Universita Degli Studi "La Sapeinza", Rome
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari
  - Struttura Complessa Ematologia - Azienda Sanitaria Locale BAT1- Presidio Ospedaliero Bisceglie-Trani, Trani
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piciocchi A, Messina M, Elia L, Vitale A, Soddu S, Testi AM, Chiaretti S, Mancini M, Albano F, Spadano A, Krampera M, Bonifacio M, Cairoli R, Vetro C, Colella F, Ferrara F, Cimino G, Bassan R, Fazi P, Vignetti M. Prognostic impact of KMT2A-AFF1-positivity in 926 BCR-ABL1-negative B-lineage acute lymphoblastic leukemia patients treated in GIMEMA clinical trials since 1996. Am J Hematol. 2021 Sep 1;96(9):E334-E338. doi: 10.1002/ajh.26253. Epub 2021 Jun 9. No abstract available. PMID 34048072